CLINICAL TRIAL: NCT01422486
Title: Phase 2 Study of Oral Ezatiostat Hydrochloride (Telintra®) in Patients With Lenalidomide (Revlimid®) Refractory or Resistant, Low to Intermediate-1 Risk, Deletion 5q Myelodysplastic Syndrome
Brief Title: Phase 2 Study of Telintra® in Deletion 5q Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study TLK199.2107 was terminated for business reasons.
Sponsor: Telik (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLK199.2107
Record Dates: First submitted 2011-08-18; First posted 2011-08-24 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Myelodysplastic Syndrome (MDS)
Keywords: Hematology; MDS; Myelodysplastic Syndrome; Low risk MDS; Intermediate-1 risk MDS; Int-1 risk MDS; Transfusion dependence; Lenalidomide refractory; Revlimid refractory; Lenalidomide resistant; Revlimid resistant; Telintra; ezatiostat; ezatiostat hydrochloride; TLK199; Glutathione; Glutathione analog; Glutathione Transferase; Glutathione Transferase P1-1 inhibitor; GST P1-1 inhibitor; Apoptosis; Differentiation; Enzyme inhibitor
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — gamma-Glu-S-BzCys-PhGly diethyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ezatiostat hydrochloride (Telintra®) (Experimental): Patients received ezatiostat at a starting dose of 2000 mg total daily dose in divided doses (1000 mg PO b.i.d.) for three weeks (21 days) on therapy followed by a one-week (7 days) off therapy rest period in four-week (28 days) treatment cycles.
  Interventions: Drug: ezatiostat hydrochloride (Telintra®)

INTERVENTIONS:
Drug: ezatiostat hydrochloride (Telintra®) — Three weeks of treatment with ezatiostat at 2000 mg per day in divided doses followed by a one week rest period in four-week treatment cycles.
  Other Names: Telintra; Telinta Tablets; Oral Telintra; ezatiostat; ezatiostat hydrochloride; oral ezatiostat

SUMMARY:
Study TLK199.2107 is a multicenter, single arm, open-label Phase 2 study of oral ezatiostat (Telintra®) in patients with lenalidomide (Revlimid®) refractory or resistant, red blood cell (RBC) transfusion-dependent, Low to Intermediate-1 IPSS risk, del5q Myelodysplastic Syndrome (MDS).

DETAILED DESCRIPTION:
Study TLK199.2107 is a multicenter, single arm, open-label Phase 2 study of oral ezatiostat (Telintra®) in patients with lenalidomide (Revlimid®) refractory or resistant, red blood cell (RBC) transfusion-dependent, Low to Intermediate-1 IPSS risk, del5q Myelodysplastic Syndrome (MDS). Independence from red blood cell transfusions, improvement in the levels of red blood cells, white blood cells, and platelets, and the response of the bone marrow were evaluated. Patients received a starting dose of 2000 mg total daily dose in divided doses (1000 mg orally twice daily for three weeks (21 days) on therapy followed by a one-week (7 days) off therapy rest period in four-week (28 days) treatment cycles. Patients continued treatment until documentation of lack of MDS response, MDS progression, unacceptable toxicity, or patient withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria:

* Primary or de Novo MDS
* Low or Intermediate-1 IPSS risk MDS
* Deletion of the 5q chromosome [del(5q) MDS]
* Refractory or resistant to lenalidomide (Revlimid)
* ECOG performance score of 0 or 1
* Documentation of significant anemia with or without additional cytopenia
* Adequate kidney and liver function
* Patients must have discontinued hematopoietic growth factors at least 3 weeks prior to study entry

Exclusion Criteria:

* Prior allogenic bone marrow transplant for MDS
* Known sensitivity to ezatiostat (injection or oral tablets)
* Prior treatment with hypomethylating agent (HMA) (e.g., azacitadine, decitabine)
* History of MDS IPSS risk score of greater than 1.0
* Pregnant or lactating women
* Any severe concurrent disease, infection or comorbidity that, in the judgement of the investigator, would make the patient inappropriate for study entry
* Oral steroids greater than 10 mg per day. Exceptions: those prescribed for other conditions (such as new adrenal failure, asthma, arthritis) or brief steroid use (such as tapered dosing for an acute non-MDS condition)
* History of hepatitis B or C, or HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Hematologic Improvement-Erythroid (HI-E) rate | At 8, 16, 24, and 32 weeks of treatment
  Hematologic Improvement response will be assessed per the IWG MDS response criteria (2006)

SECONDARY OUTCOMES:
RBC Transfusion independence (TI) rate | At 4, 8, 12, 16, 20, 24, 28 & 32 weeks of treatment
Hematologic Improvement-Neutrophil (HI-N) rate | At 8, 16, 24, & 32 weeks of treatment
  Hematologic Improvement response will be assessed per the IWG MDS response criteria (2006)
Hematologic Improvement-Platelet (HI-P) rate | At 8, 16, 24, & 32 weeks of treatment
  Hematologic Improvement response will be assessed per the IWG MDS response criteria (2006)
Unilineage, bilineage, trilineage, and overall HI response rate | 2 years
Cytogenetic response rate | 16 weeks, 48 weeks and at the time of first HI response
Duration of response | 2 years
Safety of ezatiostat in this MDS population | At 4, 8, 12, 16, 20, 24, 28 & 32 weeks of treatment
  Recording and grading of AEs using NCI-CTCAE v4.03
Evaluation of the relationship between HI-E response, gene expression profiling and response-related variables | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gail L Brown, MD, Study Director — Telik
Locations (5):
- United States (5):
  - Loyola University, Maywood, Illinois
  - SIU School of Medicine, Simmons Cancer Center, Springfield, Illinois
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Columbia University, New York, New York
  - Vanderbilt University, Nashville, Tennessee